CLINICAL TRIAL: NCT02750293
Title: The Effect of Vitamin D Supplementation on Cardiovascular Risk Factors in Subjects With Low Serum 25-hydroxyvitamin D Levels
Brief Title: The Effect of Vitamin D Supplementation on Cardiovascular Risk Factors
Acronym: D-COR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Rolf Jorde, Professor, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TromsøEndo-2013-1; 2013-003514-40 (EudraCT Number)
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; blood pressure; serum lipids; glucose metabolism; muscle function; arterial stiffness; depression; psoriasis; sleep; bone density
MeSH Terms: conditions — Vitamin D Deficiency; Depression; Psoriasis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Active Comparator): vitamin D (as a 20 000 IU capsule) will be given once a week for 4 months
  Interventions: Drug: Cholecalciferol
- placebo (Placebo Comparator): placebo capsules (identical looking to the vitamin D capsules) will be given once a week for 4 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D preparation
  Other Names: Dekristol
  Arms: cholecalciferol
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
Six-hundred subjects with vitamin D deficiency will be randomized to vitamin D 3000 IU per day versus placebo for 4 months, with effects on cardiovascular risk factors as main endpoint

DETAILED DESCRIPTION:
Vitamin D is a hormone with effects not only on the skeleton, but on most tissues in the body. Lack of vitamin D is associated with cardio-vascular disease (CVD) and type 2 diabetes, and also with risk factors for these diseases like hypertension, dyslipidemia, insulin resistance, and endothelial dysfunction. However, intervention studies with vitamin D have been inconclusive regarding diseases and risk factors. Most of these studies were done in white, Western populations in subjects fairly vitamin D sufficient, and accordingly, no benefits were to be expected. Also, in many studies the doses of vitamin D have been too low, and the studies underpowered. To firmly establish the role of vitamin D regarding CVD risk factors we will in the present study include 600 subjects with vitamin D deficiency (serum 25-hydroxyvitamin D (25(OH)D) < 30 nmol/L) and randomize to high dose vitamin D (3000 IU per day) versus placebo for four months. The subjects will be recruited based on 25(OH)D measurements in the forthcoming 7th survey in the Tromsø study where more than 20 000 subjects are expected to attend. If our hypotheses are correct and the vitamin D supplement has a positive effect, this will be of great importance not only in countries with low sun exposure, but particularly for subjects in developing countries where vitamin D deficiency is highly prevalent.

ELIGIBILITY:
Inclusion Criteria:

* participated in The 7th survey in The Tromsø study
* vitamin D deficiency

Exclusion Criteria:

* primary hyperparathyroidism
* granulomatous disease
* reduced kidney function
* systolic blood pressure > 174 mmHg
* diastolic blood pressure > 104 mmHg
* diabetes
* renal stones last 5 years
* use of solarium on regular basis
* planned holidays in tropical areas
* clinical depression
* clinical signs of vitamin D deficiency (muscle weakness)
* use of vitamin D supplements
* serious illness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure | 4 months

SECONDARY OUTCOMES:
Change from baseline in hand-grip, quadriceps and biceps muscle strength measured by hand held dynamometry . | 4 months
Change from baseline in score on Becks Depression Inventory | 4 months
Change from baseline in cognitive function evaluated with The Twelve Word Memory Test | 4 months
Change from baseline in cognitive function evaluated with The Digit Symbol Coding Test | 4 months
Change from baseline in cognitive function evaluated with The Tapping Test | 4 months
Change from baseline in arterial stiffness and endothelial function evaluated with pulse wave velocity | 4 months
Change from baseline in arterial stiffness and endothelial function evaluated with augmentation index (AIX) | 4 months
Change from baseline in arterial stiffness and endothelial function evaluated with the subendocardial viability ratio (SEVR) | 4 months
Change from baseline in number of subjects with nasal staphylococcus aureus colonization | 4 months
Change from baseline in bone mass density measured with dual energy x-ray absorptiometry (DEXA) at the lumbar spine and hip | 4 months
Change from baseline in the bone turnover marker serum type 1 procollagen (P1NP) | 4 months
Change from baseline in the bone turnover marker serum collagen type 1 cross-linked C-telopeptide (CTX-1) | 4 months
Change from baseline in serum marker of interferon-γ mediated macrophage activation | 4 months
Change from baseline in serum vitamin B6 status. | 4 months
Change from baseline in the glycosylation marker HbA1c | 4 months
Change from baseline in the glycosylation marker the receptor for advanced glycosylation end products (s-RAGE) | 4 months
Change from baseline in the glycosylation marker carboxy-methyllysine | 4 months
Change from baseline in psoriasis Activity in subjects with psoriasis evaluated with the Self-Administered Psoriasis Area Severity Index (SAPASI) | 4 months
Change from baseline in psoriasis Activity in subjects with psoriasis, evaluated with the Dermatological Life Quality Index (DLQI) | 4 months
Change from baseline in psoriasis Activity in subjects with psoriasis, evaluated with the Psoriasis Area Severity Index (PASI) | 4 months
Change from baseline in transcriptomic profile (mRNA) in adipose tissue biopsies | 4 months
Change from baseline in number of subjects with nocturnal legg cramps | 4 months
Change from baseline in sleep pattern evaluated with the Tromsø Study 7th Survey sleep pattern questionnaire | 4 months
Change from baseline in the serum total cholesterol | 4 months
Change from baseline in the serum HDL-cholesterol | 4 months
Change from baseline in the serum LDL-cholesterol | 4 months
Change from baseline in the serum triglycerides | 4 months
Change from baseline in the serum Apolipoprotein A1 | 4 months
Change from baseline in the serum Apolipoprotein B, | 4 months
Change from baseline in insulin resistance evaluated with the homeostasis model assessment (HOMA) index based on fasting serum glucose and serum insulin | 4 months
Change from baseline in proteomic profile with relative quantification in adipose tissue biopsies with the use of Liquid chromatography mass spectrometry Technology (LC-MS/MS) | 4 months
Change from baseline in metabolomic profile with relative quantification in adipose tissue biopsies with the use of Liquid chromatography mass spectrometry Technology (LC-MS/MS) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Derived] Jorde R, Kubiak J, Svartberg J, Fuskevag OM, Figenschau Y, Martinaityte I, Grimnes G. Vitamin D supplementation has no effect on cognitive performance after four months in mid-aged and older subjects. J Neurol Sci. 2019 Jan 15;396:165-171. doi: 10.1016/j.jns.2018.11.020. Epub 2018 Nov 17. PMID 30472553